CLINICAL TRIAL: NCT07081607
Title: An Open-label, Single-arm Study Evaluating the Safety and Efficacy of Golidocitinib Combined With Azacitidine and Chidamide in Patients With Peripheral T-cell Lymphoma.
Brief Title: Golidocitinib With Azacitidine and Chidamide in Patients With Peripheral T-cell Lymphoma.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director，Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-chemofree
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Peripheral T-Cell Lymphoma, Not Classified
Keywords: Golidocitinib; Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golidocitinib with azacytidine and chidamide (Experimental)
  Interventions: Drug: golidocitinib with azacytidine and chidamide

INTERVENTIONS:
Drug: golidocitinib with azacytidine and chidamide — In Phase I, a "3+3" dose-escalation design will be adopted to enroll 3 to 12 participants, exploring the recommended Phase II dose (RP2D) at two dose levels of golidocitinib: 150 mg every other day (QOD) and 150 mg once daily (QD).
  In Phase II, we aim to evaluate the efficacy and safety of golidocitinib RP2D po in combination with chidamide 20mg biw po and azacytidine 100mg d1-7, SC in patients with peripheral T-cell lymphoma

SUMMARY:
In decades, the outcome of patients with peripherial T-cell lymphomas is dismal, especially in relapsed or refractory population. After failure to the frontline treatment, patients have limited treatment options and elderly population usually have no chance to undergo transplantation due to age or comorbidity, etc. Golidocitinib and chidamide were approved in treating r/r PTCL in China, while azacytidine has been demonstrated its anti-tumor activity in PTCL as well.

This study aims to explore the efficacy and safety of golidocitinib combined with azacytidine and chidamide in the patients with peripheral T-cell lymphoma who are eligible for intensive chemotherapy or transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed peripheral T-cell lymphoma;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2;
3. Expected survival of ≥12 weeks;
4. Measurable disease lesions;
5. Any conditions considered ineligible for intenvive chemotherapy, including but not limted to age > 60 years, at least one comorbidity scored 3 points, or more than 4 comorbidities scored 2 points each according to the CIRS scale;
6. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to and adhere to effective contraceptive measures during the treatment period and for 180 days after the last dose of the study drug;
7. Participants must voluntarily join the study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up assessments.

Exclusion Criteria:

1. Involvement of the central nervous system (CNS);
2. History of malignancies except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix;
3. Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
4. Left ventricular ejection fraction<50%
5. Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

   * Neutrophils<1.5×10^9/L
   * Platelets<75×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement)
   * ALT or AST is 2 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.
   * Creatinine is 1.5 times higher than the ULN.
6. HIV-infected patients
7. Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
8. Pregnant or lactation
9. Require treatment with strong/moderate CYP3A inhibitors or inducers.
10. Inability to swallow capsules or presence of diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, post-bariatric surgery, inflammatory bowel disease and complete or incomplete intestinal obstruction
11. Other medical conditions determined by the researchers that may affect the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 21 days) through study completion, an average of 1 year
  Percentage of participants with complete response or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off(up to approximately 3 years)
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Complete Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 21 days) through study completion, an average of 1 year.
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of Response | Baseline up to data cut-off(up to approximately 3 years)
  Applicable to complete or partial response participants. DoR was defined as the time from the first documented date of complete or partial response until the date of the disease progression or death from any causes.
Overall survival | Baseline up to data cut-off(up to approximately 3 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

IPD SHARING:
Plan to Share IPD: No